CLINICAL TRIAL: NCT03472092
Title: Distinct Mechanisms of Cognitive Behavioral Therapy Effects in Youth With Migraine & Dissecting Neural Mechanisms Supporting Mind and Body Approaches to Pain Reduction in Youth With Migraine
Brief Title: Mind and Body Approaches to Pain Reduction in Youth With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CAP Imaging Study I-II; R01NS101321 (NIH); R01AT010171 (NIH)
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Headache, Migraine; Migraine; Migraine Disorders; Headache
Keywords: headache; migraine; cognitive behavioral therapy; amitriptyline; functional magnetic resonance imaging; conditioned pain modulation; brain connectivity; pediatrics
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Cognitive Behavioral Therapy; Coping Skills; Amitriptyline

STUDY DESIGN:
Intervention Model Description: Mechanistic/basic science project seeking to identify the neural mechanisms by which youth with migraine improve in response to preventive treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Behavioral therapy assignment is known to the treating therapist/care provider. Placebo and amitriptyline are double blinded. Participant will be aware they are either assigned to behavioral or pill therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cognitive Behavioral Therapy (CBT) (Experimental): Cognitive Behavioral Therapy (CBT) is a mind and body based intervention using education on gate control theory of pain, behavioral strategies such as muscle relaxation and activity pacing, and cognitive strategies including distraction, problem solving, and using calming self-statements.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Placebo (Placebo Comparator): The placebo pill will be administered once a day at home, to be taken by mouth.
  Interventions: Drug: Placebo
- Amitriptyline (Active Comparator): Amitriptyline will be administered once a day at home, to be taken by mouth. Dosage will be weight-based.
  Interventions: Drug: Amitriptyline
- Biofeedback-Assisted Relaxation Training (BART) (Active Comparator): Biofeedback-Assisted Relaxation Training (BART) is a mind and body based intervention that focuses specifically on mind and body techniques such as deep breathing, muscle relaxation, and guided imagery skills to manage pain.
  Interventions: Behavioral: Biofeedback-Assisted Relaxation Training (BART)
- Cognitive Retraining (CR) (Active Comparator): Cognitive Retraining (CR) is a mind and body based intervention that focuses on the use of tests of evidence and other cognitive strategies such as positive coping statements and pleasant activities and mindfulness to manage pain.
  Interventions: Behavioral: Cognitive Reappraisal Training (CR)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — This intervention will consist of 8 weekly sessions. The duration of each session is about 45 minutes and will be led by a psychologist/therapist using a manualized protocol. About half of the sessions will be conducted in person and the remaining sessions will be offered via telehealth (Skype or phone).
  Other Names: CBT; coping skills; mind body relaxation
  Arms: Cognitive Behavioral Therapy (CBT)
Drug: Placebo — The placebo pill will be administered once a day at home for 8 weeks, to be taken by mouth with or without food under the supervision of the participant's parent or guardian. To maintain blinding, all participants will receive 1 matching capsule as a daily dose to be taken each evening during the study.
  Other Names: Placebo Oral Capsule
  Arms: Placebo
Drug: Amitriptyline — Amitriptyline will be administered once a day at home for 8 weeks, to be taken by mouth with or without food under the supervision of the participant's parent or guardian. To maintain blinding, all participants will receive 1 matching capsule as a daily dose to be taken each evening during the study. For this study, a dose of 0.25 mg/kg/day will be provided for the 1st 2 weeks, followed by a dose of 0.5 mg/kg/day for 2 weeks, 0.75 mg/kg/day for 2 weeks and a maximum dose of 1.0 mg/kg/day for 2 weeks based on tolerability. Participants experiencing tolerability issues, may be held a current dose rather than titrated to the next dosage if deemed appropriate by the study doctor.
  Other Names: Elavil
  Arms: Amitriptyline
Behavioral: Biofeedback-Assisted Relaxation Training (BART) — This intervention will consist of 8 weekly sessions. The duration of each session is about 45 minutes and will be led by a psychologist/therapist using a manualized protocol. About half of the sessions will be conducted in person and the remaining sessions will be offered via telehealth (Skype or phone).
  Arms: Biofeedback-Assisted Relaxation Training (BART)
Behavioral: Cognitive Reappraisal Training (CR) — This intervention will consist of 8 weekly sessions. The duration of each session is about 45 minutes and will be led by a psychologist/therapist using a manualized protocol. About half of the sessions will be conducted in person and the remaining sessions will be offered via telehealth (Skype or phone).
  Arms: Cognitive Retraining (CR)

SUMMARY:
The overarching objective of this protocol is to identify and understand the neural and pain processing mechanisms by which youth with migraine improve in response to preventive treatment. The study design of this mechanistic investigation includes functional magnetic resonance imaging (fMRI), daily headache diaries, assessment of conditioned pain modulation via quantitative sensory testing, and validated psychometric assessments before and after the delivery of one of five treatments over an 8 week period [cognitive behavioral therapy (CBT), biofeedback-assisted relaxation training (BART) and cognitive reappraisal (CR) training, amitriptyline, and placebo]. We are examining both distinct and common pathways that may help explain the response to various preventive treatments, as well as potential predictors of outcome.

DETAILED DESCRIPTION:
Pediatric migraine is a prevalent disorder that results in significant pain and disability for children and adolescents. Despite the prevalence and cost, commonly used pharmacologic treatments to treat pediatric migraine have limited evidence of efficacy over placebo in preventing migraine in youth. In our prior research, published in NEJM (Trial of Amitriptyline, Topiramate, and Placebo for Pediatric Migraine. N Engl J Med. 2017;376(2):115-124),we have shown in a large, national, multicenter trial that the most widely used conventional preventive medications, amitriptyline (AMI) and topiramate, are no more effective than placebo. Psychological therapies for pediatric headache (in particular, cognitive behavioral therapy [CBT]) result in better outcomes than control conditions by effectively reducing headache days and disability in children and adolescents with migraine. Our own work indicates that youth receiving combined CBT plus amitriptyline (AMI, the most widely used migraine prophylactic in youth) had greater reductions in headache days and disability than a group receiving education control plus AMI. Specifically, we found that CBT combined with AMI improved outcomes for about 2 out of 3 pediatric chronic migraineurs (ages 10-17). Reduction in headache days by ≥ 50% was seen within the first 8 weeks of this 5-month trial (Powers SW, Kashikar-Zuck SM, Allen JR, et al. Cognitive behavioral therapy plus amitriptyline for chronic migraine in children and adolescents: a randomized clinical trial. JAMA. 2013;310(24):2622-2630).

Despite this evidence of efficacy, the mechanisms supporting CBT for migraine remain poorly understood. This lack of mechanistic understanding leaves patients, providers, and payers reluctant to promote CBT as a primary treatment modality. Moreover, opportunities to optimize and individualize CBT remain unrealized because of limited basic understanding by which different components of CBT exert their effects. Little remains known about the specific brain mechanisms by which CBT reduces pain. Therefore, it is critical that we understand how and why CBT may improve headache outcomes in contrast to pill-taking treatments, specifically placebo. Brain imaging and quantitative sensory testing are novel tools to investigate possible mechanisms of CBT, placebo, and medication. In addition understanding the components of CBT and how they may work at the brain and pain processing levels is important. As such, two broad components of CBT represent clear targets for investigation: relaxation and cognitive reappraisal.

Evolving consensus in the pain community and at a national level suggests that examining biological mechanisms of how mind and body approaches lead to benefits for patients will advance care, improve outcomes, and legitimize non-pharmacological treatment for pediatric chronic pain. As such, this mechanistic/basic science study seeks to identify the neural mechanisms by which youth with migraine improve in response to preventive treatment. Pediatric medical and behavioral clinicians can use mechanistic insights from this study to provide patients and families with a stronger rationale for treatment, thereby decreasing stigma and increasing confidence in and commitment to the care plan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Migraine with or without aura or chronic migraine that meets the International Classification of Headache Disorders, 3rd Edition (beta) (ICHD-3b) criteria
* Frequency: Headache frequency based upon prospective headache diary of 28 days must be ≥ 8 and ≤ 28
* PedMIDAS: PedMIDAS Disability Score > 10, indicating at least mild disruption in daily activities and < 140, indicating extreme disability that may require more comprehensive, multi-component therapy
* English speaking: able to complete interviews and questionnaires in English

Exclusion Criteria:

* Continuous migraine defined as an unrelenting headache for a 28 day period
* Weight less than 30 kg or greater than 120 kg, or weight/size incompatible with magnetic resonance imaging (MRI) scanner
* Must agree not to take non-specific acute medication, such as nonsteroidal anti-inflammatory drugs (NSAIDS) (e.g., ibuprofen), more than 3 times per week, or migraine specific acute medications, such as triptans, more than 6 times per month
* No current prophylactic anti-migraine medication within a period equivalent to < 5 half-lives of that medication before entering the screening phase, and agree to not begin a migraine prevention medication during the study period
* Current use of the following medications/products: opioids, antipsychotics, antimanics, barbiturates, benzodiazepines, muscle relaxants, sedatives, tramadol, nutraceuticals
* Known history of allergic reaction or anaphylaxis to amitriptyline
* Abnormal findings on electrocardiogram (ECG) at baseline, particularly lengthening of the QT interval ≥ 450 msec
* Orthodontic braces, metallic or electronic implants, or other metal objects in the body which obscure or interfere with the MRI, or pose a risk from heating, movement, or malfunction in the MRI environment
* Claustrophobia
* Youth who are pregnant, or those who are sexually active and not using a medically accepted form of contraception (barrier or hormonal methods)
* Diagnosis of epilepsy or other neurological diseases
* Inability to learn how to swallow pills using behavioral techniques (if indicated)
* Present psychiatric disease as defined by the Diagnostic and Statistical Manual (DSM) IV (e.g. psychosis, bipolar disorder, major depression, generalized anxiety disorder), alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, attention deficit hyperactivity disorder (ADHD), or mental retardation) that, in the opinion of the investigator, would interfere with adherence to study requirements or safe participation in the study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in functional resonance imaging (fMRI) | baseline and post treatment (8 weeks post randomization)
  For each study group, changes in distinct neural mechanisms of the brain will be compared to between baseline and post treatment (8 weeks). For each study group, the primary endpoint will be examine changes in brain connectivity and activation.
Conditioned pain modulation as measured in a standard protocol using quantitative sensory testing. Employed as a predictor of headache day change in the study analytic plan | baseline and post treatment (8 weeks post randomization)
  Conditioned pain modulation as measured by quantitative sensory testing will be established for each participant. This measure involves testing pain tolerance of pressure and cold pain stimuli in a controlled manner using a standard protocol. Baseline levels of CPM for each study group will be used to predict headache day reduction for each study group. The hypothesis to be tested is that low efficiency of CPM will be differentially predictive of headache reductions following CBT in relation to other study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Powers, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Robert Coghill, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03472092/ICF_000.pdf